CLINICAL TRIAL: NCT06241742
Title: A Phase-2 Study to Evaluate the Ability of HT-6184 to Attenuate Diagnostic Biomarkers of Post-procedure Acute Inflammation and Manage Pain Following Third Molar Extraction
Brief Title: Evaluating Ability of HT-6184 to Reduce Inflammation and Pain After Third Molar Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Halia Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HT-6184-PIR-001
Record Dates: First submitted 2024-01-15; First posted 2024-02-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pain
Keywords: third molar extraction; inflammation; biomarkers
MeSH Terms: conditions — Pain; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HT-6184 Treatment Arm (Active Comparator)
  Interventions: Drug: HT-6184
- HT-6184 Placebo (Placebo Comparator)
  Interventions: Drug: HT-6184 Placebo

INTERVENTIONS:
Drug: HT-6184 — Single, oral dose of HT-6184
  Arms: HT-6184 Treatment Arm
Drug: HT-6184 Placebo — Single, oral dose of placebo
  Arms: HT-6184 Placebo

SUMMARY:
The goal of this clinical trial is to test the ability of HT-6184 to decrease inflammation and pain in patients after third molar removal.

The main question it aims to answer are:

* Does HT-6184 decrease inflammation in patients after third molar removal?
* Does HT-6184 decrease pain in patients after third molar removal?

Participants will be asked to do the following during the clinical trial:

* Take a single oral dose of HT-6184 or placebo
* Allow a oral surgeon remove their third molar teeth
* Blood draws on 5 occurrences
* Rate their pain intensity
* Attend two follow-up appointments on day 1 and day 2 after third molar removal
* Participate in one follow-up phone call 5-7 days after third molar removal

ELIGIBILITY:
Inclusion Criteria:

* The candidate is 18 years of age or older, capable of understanding and providing written informed consent to participate and willing to comply with study procedures including providing a blood sample to be saved for potential pharmacokinetic and/or genetic analysis.
* The candidate, for any reason, requires surgical extraction of two or more third molars of which at least one is partially or fully impacted in mandibular bone.
* The candidate is postmenopausal, surgically sterile or agrees to use an effective and medically acceptable method of contraception for 1 week after his or her last dose of study drug.
* If female with child-bearing potential, the candidate must have a negative pregnancy test at screening and pre-surgery on the day of surgery.

Exclusion Criteria:

* The candidate typically or on average consumes more than one alcoholic beverage per day.
* The candidate is pregnant or nursing.
* The candidate has received an investigational drug or used an experimental medical device within 30 days prior to screening.
* The candidate has donated 1 or more pints of blood within 8 weeks prior to screening.
* The candidate has any hypersensitivity to components of the HT-6184/placebo formulations or the protocol-specified analgesic rescue medication, aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs).
* The candidate has any contraindication to oral surgery or any serious or major medical problems that, in the investigator's opinion, may compromise the safety or the candidate or interfere with the interpretation of study results
* The candidate has taken acetaminophen, NSAIDs (including aspirin) or other medications for pain within 72 hours of the surgical procedure.
* The candidate has any abnormal laboratory value or physical finding that, in the opinion of the investigator, may compromise the individual's safety, interfere with interpretation of the study results, or be indicative of an underlying disease state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in serum C-reactive protein levels from pre-dose | Up to 54 hours post surgery
Incidence of adverse events | Up to 7 days post surgery
  Severity of AEs will be judged according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Incidence of serious adverse events | Up to 7 days post surgery
  Severity of AEs will be judged according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Area under the categorical pain intensity-by-time curve (AUCs) | Up to 8 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Halia Study Director, Study Director — Halia Therapeutics
Locations (1):
- CenExel JBR, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No